CLINICAL TRIAL: NCT07283653
Title: Dissemination and Implementation of DIGEST™ as an Evidence-based Measurement Tool for Dysphagia: A Randomized Implementation Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-1270
Record Dates: First submitted 2025-12-10; First posted 2025-12-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: DIGEST; Evidence Based Measurement; Dysphagia; Randomized Implementation
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm 1 (Experimental): The control arm will receive no active implementation strategy.
  Interventions: Other: No intervention
- Training Arm 2 (Experimental): Represents a low intensity implementation strategy solely using the DIGEST training program as the intervention.
  Interventions: Other: DIGEST Training Program
- Training + Practice Facilitation Arm 3 (Experimental): Represents a higher intensity strategy using the same training program plus practice facilitation.
  Interventions: Other: DIGEST Training + Practice Facilitation

INTERVENTIONS:
Other: No intervention — receive no active implementation
  Arms: Control Arm 1
Other: DIGEST Training Program — Investigator led training program
  Arms: Training Arm 2
Other: DIGEST Training + Practice Facilitation — Training plus practice facilitation
  Arms: Training + Practice Facilitation Arm 3

SUMMARY:
To improve swallowing outcomes in cancer through clinical implementation of the Dynamic Imaging Grade of Swallowing Toxicity (DIGEST™) as an evidence-based practice (EBP) tool to grade pharyngeal dysphagia (difficulty swallowing) as a toxicity of cancer.

DETAILED DESCRIPTION:
Primary Objective Assess the impact of implementation strategies on clinical adoption (reach) of DIGEST for oncology MBS studies.

Secondary Objective Assess the impact of implementation strategies on the fidelity (reliability) of DIGEST adoption for oncology MBS studies

ELIGIBILITY:
Inclusion Criteria:

1. A hospital or clinic affiliated with the Veteran's Affairs system, University of Wisconsin system, or Ohio State University system.
2. A minimum average of 10 Modified Barium Swallow (MBS) procedures per month in oncology patients in preceding year.
3. MBS imaging files are recorded and archived as a routine procedure (and accessible to researchers).

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Adoption of DIGEST in routine clinical documentation for oncology MBS studies | Through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kate Hutcheson, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://mdanderson.org